CLINICAL TRIAL: NCT05028790
Title: Evaluating Contact Lens Optics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David A Berntsen, OD PhD (Other)
Responsible Party: Sponsor-Investigator, David A Berntsen, OD PhD, Associate Professor, University of Houston
Organization: University of Houston (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY00002545
Record Dates: First submitted 2021-08-25; First posted 2021-08-31 (Actual); Results first posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants were masked to the order in which they wore contact lenses
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Single vision soft contact lens first, then multifocal soft contact lens (Experimental): Participants wore the single vision soft contact lens first, then a multifocal soft contact lens
  Interventions: Device: Single vision contact lens; Device: Multifocal contact lens
- Multifocal soft contact lens first, then single vision soft contact lens (Experimental): Participants wore the multifocal soft contact lens first, then the single vision soft contact lens
  Interventions: Device: Single vision contact lens; Device: Multifocal contact lens

INTERVENTIONS:
Device: Single vision contact lens — Participants will wear a single vision soft contact lens during the study visit
  Other Names: comfilcon A
Device: Multifocal contact lens — Participants will wear a multifocal soft contact lens during the study visit
  Other Names: comfilcon A

SUMMARY:
This study will evaluate changes in refractive error and visual performance between a single vision soft contact lens and multifocal soft contact lens

ELIGIBILITY:
Inclusion Criteria:

* Able to read and understand the informed consent document
* 18 to 39 years of age (inclusive)
* Best corrected visual acuity of 20/25 or better in the right eye
* Refractive error from -1.00D to -6.00D with astigmatism less than or equal to -1.00D in the right eye (corneal plane)

Exclusion Criteria:

* Any ocular or systemic conditions affecting vision, refraction, or the ability to wear a soft contact lens
* History of ocular trauma or surgery causing abnormal or distorted vision
* Current Rigid Gas Permeable (RGP) contact lens wearers
* Unwilling to have contact lens fit photographed
* Pregnant and/or lactating females, by self-report

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-27 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Berntsen, OD, PhD, Principal Investigator — University of Houston College of Optometry
Locations (1):
- University of Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Vision Soft Contact Lens First, Then Multifocal Soft Contact Lens: Participants wore the single vision soft contact lens first, then the multifocal soft contact lens
Period: First Intervention (40 Mins)
Arm/Group | Single Vision Soft Contact Lens First, Then Multifocal Soft Contact Lens | Multifocal Soft Contact Lens First, Then Single Vision Soft Contact Lens
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0
Period: Washout (5 Mins)
Arm/Group | Single Vision Soft Contact Lens First, Then Multifocal Soft Contact Lens | Multifocal Soft Contact Lens First, Then Single Vision Soft Contact Lens
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0
Period: Second Intervention (40 Mins)
Arm/Group | Single Vision Soft Contact Lens First, Then Multifocal Soft Contact Lens | Multifocal Soft Contact Lens First, Then Single Vision Soft Contact Lens
Started | 9 | 7
Completed | 9 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Vision Soft Contact Lens First, Then Multifocal Soft Contact Lens | Multifocal Soft Contact Lens First, Then Single Vision Soft Contact Lens | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.11 (1.83) | 24 (1.15) | 24.63 (1.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 7 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 0 | 3
  White | 4 | 4 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Visual Performance
Description: Low contrast visual acuity was measured for each participant while wearing each of the two lenses
Time Frame: Through completion of study visit, an average of 2.5 hours
Measure: Mean (Standard Deviation); unit: logMAR
Groups:
- Single Vision Contact Lens: Low contrast visual acuity measured while participants were wearing the single vision soft contact lens
- Multifocal Contact Lens: Spherical equivalent refractive error measured while participants were wearing the multifocal soft contact lens
Arm/Group | Single Vision Contact Lens | Multifocal Contact Lens
Number analyzed (Participants) | 9 | 7
logMAR | 0.23 (0.08) | 0.38 (0.12)

2. Secondary Outcome: Spherical Equivalent Refractive Error On-axis
Description: Refraction was measured after cycloplegia with two drops of 1% tropicamide hydrochloride. Spherical equivalent refractive error was then measured 3 times with an aberrometer and averaged.
Time Frame: Through completion of study visit, an average of 2.5 hours
Measure: Mean (Standard Deviation); unit: D
Groups:
- Single Vision Soft Contact Lens: Spherical equivalent refractive error measured while participants were wearing the single vision soft contact lens
- Multifocal Soft Contact Lens: Spherical equivalent refractive error measured while participants were wearing the multifocal soft contact lens
Arm/Group | Single Vision Soft Contact Lens | Multifocal Soft Contact Lens
Number analyzed (Participants) | 16 | 16
D | 0.61 (0.46) | 0.17 (0.44)

3. Secondary Outcome: Spherical Equivalent Refractive Error at 30 Degrees Temporal Retina
Description: Cycloplegic spherical equivalent refractive error was measured 3 times with an aberrometer and averaged.
Time Frame: Through completion of study visit, an average of 2.5 hours
Measure: Mean (Standard Deviation); unit: D
Groups:
- Single Vision Contact Lens: Spherical equivalent refractive error measured while participants were wearing the single vision soft contact lens
Arm/Group | Single Vision Contact Lens | Multifocal Contact Lens
Number analyzed (Participants) | 16 | 16
D | 0.68 (1.03) | -1.20 (1)

4. Secondary Outcome: Spherical Equivalent Refractive Error at 20 Degrees Temporal Retina
Description: Cycloplegic spherical equivalent refractive error was measured 3 times with an aberrometer and averaged.
Time Frame: Through completion of study visit, an average of 2.5 hours
Measure: Mean (Standard Deviation); unit: D
Arm/Group | Single Vision Contact Lens | Multifocal Contact Lens
Number analyzed (Participants) | 16 | 16
D | 0.52 (0.68) | -1.30 (0.44)

5. Secondary Outcome: Spherical Equivalent Refractive Error at 20 Degrees Nasal Retina
Description: Cycloplegic spherical equivalent refractive error was measured 3 times with an aberrometer and averaged.
Time Frame: Through completion of study visit, an average of 2.5 hours
Measure: Mean (Standard Deviation); unit: D
Arm/Group | Single Vision Contact Lens | Multifocal Contact Lens
Number analyzed (Participants) | 16 | 16
D | 0.67 (0.58) | -0.17 (0.57)

6. Secondary Outcome: Spherical Equivalent Refractive Error at 30 Degrees Nasal Retina
Description: Cycloplegic spherical equivalent refractive error was measured 3 times with an aberrometer and averaged.
Time Frame: Through completion of study visit, an average of 2.5 hours
Measure: Mean (Standard Deviation); unit: D
Arm/Group | Single Vision Contact Lens | Multifocal Contact Lens
Number analyzed (Participants) | 16 | 16
D | 0.77 (0.70) | -0.75 (0.60)

ADVERSE EVENTS:
Time Frame: 2.5 hours
Groups:
- Single Vision Contact Lens: Participants wore a single vision contact lens
- Multifocal Contact Lens: Participants wore a multifocal contact lens
Arm/Group | Single Vision Contact Lens | Multifocal Contact Lens
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/7
Other Adverse Events (participants affected / at risk) | 0/9 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT05028790/Prot_SAP_002.pdf
  • Informed Consent Form (2020-10-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT05028790/ICF_003.pdf